CLINICAL TRIAL: NCT06635109
Title: Investigation of the Effect of Different Severities of Carpal Tunnel Syndrome on Activity and Participation
Brief Title: Investigating the Effect of Carpal Tunnel Syndrome on Activity and Participation
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Phd, Kutahya Health Sciences University
Other Study IDs: 2024-a
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild carpal tunnel syndrome
- Middle carpal tunnel syndrome
- Severe carpal tunnel syndrome

SUMMARY:
The aim of our study was to examine the effect of different severities of Carpal Tunnel Syndrome on activity and participation within the framework of the International Classification of Functioning, Disability and Health (ICF).

DETAILED DESCRIPTION:
Individuals between the ages of 18-65 who were diagnosed with CTS in the dominant hand and who volunteered to participate in the study were included. SF-36, Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH), Michigan Hand Outcomes Questionnaire and Boston Carpal Tunnel Questionnaire - Functional Status Scale will be used to assess activity and participation. The questionnaires will be filled out via Google Forms. Shapiro-Wilk test will be performed to determine the distribution of the data. Whether the dependent variables differ between groups will be analysed by One-way ANOVA (continuous). For significant F-test, an additional investigation of differences between groups will be performed with Gabriel's post hoc procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CTS in the dominant hand
* Being between the ages of 18-65
* Volunteering to participate in the study

Exclusion Criteria:

* Having systemic inflammatory disease
* Having a disease that may cause polyneuropathy such as diabetes mellitus
* Having a pacemaker
* Having a disease affecting the central nervous system
* Having cervical radiculopathy
* History of previous operation or local steroid injection due to CTS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 18-65 who were diagnosed with CTS in the dominant hand and who volunteered to participate in the study were included.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Short Form - 36 Quality of Life Questionnaire (SF-36) | 15 minutes
  SF-36 is a health-related quality of life questionnaire consisting of 8 scales (physical functioning, role limitations due to physical health problems, pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, mental health). Responses to items are converted into scale scores from 0 (worst health) to 100 (best health).
Quick Disabilities of the Arm, Shoulder, and Hand (Q-DASH) | 10 minutes
  Each question in the scale is scored between 1 and 5. The results range from 0 (no difficulty or symptoms) to 100 (no activity or very severe symptoms).
Michigan Hand Questionnaire (MHQ) | 15 minutes
  The Michigan Hand Questionnaire (MHQ) is a hand-specific questionnaire that measures the health status of patients with acute and chronic hand disorders. The MHQ is an outcome tool consisting of 37 questions and 6 domains: (1) overall hand function, (2) activities of daily living, (3) pain, (4) work performance, (5) aesthetics, and (6) patient satisfaction with function. Each domain is scored using an unweighted method by summing the responses on each scale (1 to 5) and normalising the scores to a scale from 0 to 100. A lower score indicates more severe disability, other than pain. The final score is obtained by averaging the six scores after inverting the pain score.
Boston Carpal Tunnel Questionnaire - Functional Status Scale | 5 minutes
  It is an 8-item questionnaire used to assess the functional status of patients with CTS. Each item is scored from 1 to 5. Scores range from 1 (no functional deficit) to 5 (worst possible function). The patient's functional status score is the average of all 8 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)